CLINICAL TRIAL: NCT00684099
Title: A Phase I/II Study Of The Docetaxel/Pemetrexed Combination As First Line Treatment In Patients With Advanced/Metastatic NSCLC
Brief Title: Docetaxel/Pemetrexed as 1st Line Treatment in Patients With Non Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hellenic Oncology Research Group (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: V.Georgoulias, University Hospital of Crete
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT/05.18
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2009-12

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC; Pemetrexed; Docetaxel
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Docetaxel; Drug: Pemetrexed

INTERVENTIONS:
Drug: Docetaxel — Docetaxel at starting dose of 65 mg/m2 IV on day 1 every 3 weeks for a total of 6 cycles
  Other Names: Taxotere
Drug: Pemetrexed — Pemetrexed at starting dose of 400 mg/m2 IV on day 1 every 3 weeks for a total of 6 cycles
  Other Names: Alimta

SUMMARY:
This trial will determine the maximum tolerated dose the recommended phase II dose and the efficacy of this combination in locally advanced or metastatic NSCLC patients

DETAILED DESCRIPTION:
Docetaxel as single-agent therapy (100 mg/m2 and 75 mg/m2, every 3 weeks) produces response rates of 26% to 54%. Docetaxel has proven superior compared to best supportive care (BSC) in chemotherapy-naïve as well as in platinum pretreated patients. In addition, docetaxel is active in cisplatin refractory or resistant patients, producing responses ranging from 18% to 25%, implying a lack of cross-resistance between docetaxel and cisplatin, probably due to their different mechanisms of action. Furthermore, docetaxel is associated with significant prolongation of survival when administered as second line therapy, in pretreated patients with advanced NSCLC. Phase II studies of pemetrexed in previously untreated patients with NSCLC have demonstrated single agent response rates of 17% to 23%. A phase II study of pemetrexed in patients with advanced NSCLC, who had progressed during or within 3 months of completing first-line chemotherapy, demonstrated a response rate of 8.9% and median survival time of 5.7 months. Multivariate analysis established an association between an increased risk of severe pemetrexed toxicity and elevated homocysteine (folate and/or B12 vitamin deficiency marker) levels. Since December 1999, all pemetrexed-treated patients are required to receive folic acid and Vitamin B12. A recently reported phase III study compared pemetrexed with docetaxel as 2nd line therapy in patients with advanced NSCLC. Treatment with pemetrexed resulted in clinically equivalent efficacy outcomes, but with significantly fewer side effects compared with docetaxel.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed inoperable (stage IIIB-IV) NSCLC. A block of Formaline Fixed Parafine Embedded tissue representative for the primary diagnosis should be available for genomic analysis (phase II part)
* Written informed consent
* Prior chemotherapy with platinum compounds in association with or without taxanes (phase I part)
* Previously untreated with docetaxel and pemetrexed (phase II part)
* Bidimensionally, non-irradiated measurable disease (according to RECIST criteria) (phase II)
* Age ≥18 years
* World Health Organization (WHO) performance status (PS) 0-2
* Life expectancy of at least 12 weeks
* Serum bilirubin less than 1.5 times the upper normal limit (UNL)
* AST and ALT less than 2.5 times the UNL in the absence of demonstrable liver metastases, or less than 5 times the UNL in the presence of liver metastases.
* Serum creatinine less than 1.5 times the UNL
* Neutrophil count more than 1.5x 109 /L
* Platelet count more than 100x 109 /L

Exclusion Criteria:

* Other co-existing malignancies or malignancies diagnosed within the last 5 years (with the exception of basal cell carcinoma or cervical cancer in situ)
* Any evidence of severe uncontrolled concomitant disease (in the opinion of the investigator)
* Any unresolved chronic toxicity greater than CTC grade 2 from previous anticancer therapy
* Patients with unstable central nervous system metastases
* Malnutrition (loss of ≥ 20% of the original body weight)
* Performance status: 4
* Psychiatric illness or social situation that would preclude study compliance
* Pregnant or lactating women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2006-05; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of Dose Limited Toxicity and Maximum Tolerated Dose for the docetaxel/pemetrexed doublet | 2 years

SECONDARY OUTCOMES:
Response rate for the docetaxel/pemetrexed doublet | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Vassilis Georgoulias, MD, Principal Investigator — University Hospital of Crete; Athanasios Kotsakis, MD, Principal Investigator — University Hospital of Crete
Locations (8):
- Greece (8):
  - University General Hospital of Alexandroupolis, Dep of Medical Oncology, Alexandroupoli
  - "IASO" General Hospital of Athnes, Dep of Medical Oncology, Athens
  - "Laikon" General Hospital, Medical Oncology Unit, Propedeutic Dep of Internal Medicine, Athens
  - Air Forces Military Hospital, Dep of Medical Oncology, Athens
  - Sismanogleio General Hospital, 1st, 2nd Dep of Pulmonary Diseases, Athens
  - Sotiria" General Hospital, 1st Dep of Pulmonary Diseases, Athens
  - "Diabalkaniko" Hospital of Thessaloniki, Thessaloniki
  - "Theagenion" Anticancer Hospital of Thessaloniki, Thessaloniki

REFERENCES:
- [Derived] Kotsakis A, Agelaki S, Vardakis N, Stathopoulos G, Vamvakas L, Kalykaki A, Kentepozidis N, Kontopodis E, Sfakiotaki G, Mavroudis D, Georgoulias V. A dose-escalation study of pemetrexed and docetaxel in non-small-cell lung cancer. Cancer Chemother Pharmacol. 2011 Aug;68(2):415-22. doi: 10.1007/s00280-010-1508-5. Epub 2010 Nov 11. PMID 21069335